CLINICAL TRIAL: NCT04204200
Title: Prevention of Complex Regional Pain Syndrome Using Liposomal Encapsulated Vitamin C in Programmed Knee Surgery; A Prospective Randomized Trial
Brief Title: "Liposomal Encapsulated Vitamin C in Complex Regional Pain Syndrome"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Ham (Other)
Responsible Party: Principal Investigator, Jean-François Cazeneuve, Surgeon, MD, Centre Hospitalier de Ham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHHam
Record Dates: First submitted 2019-12-13; First posted 2019-12-18 (Actual); Results first posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Complex Regional Pain Syndrome I of Lower Limb

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Allocated to conventional vitamin C (n= 22) (Active Comparator): * Received allocated conventional vitamin C (n= 22)
  * Did not receive allocated conventional vitamin C (n= 0)
  Interventions: Dietary Supplement: standard vitamin C
- Allocated to liposomal vitamin C (n= 22) (Active Comparator): * Received allocated liposomal vitamin C (n= 22)
  * Did not receive allocated liposomal vitamin C (n= 0)
  Interventions: Dietary Supplement: liposomal vitamin C
- Allocated to placebo (n= 22) (Placebo Comparator): * Received allocated intervention (n= 22)
  * Did not receive allocated intervention (n= 0)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: liposomal vitamin C — The intake of liposomal vitamin C at 500 mg, in the morning and evening, one week before surgery, one during the day of surgery and lastly, during the first 21 post operation days.
  Arms: Allocated to liposomal vitamin C (n= 22)
Dietary Supplement: standard vitamin C — The intake of traditional vitamin C with a daily intake of 500 mg in the morning and evening for 28 days (starting 7 days before the operative procedure, on the day of the surgery and ending twenty-one days after surgery).
  Arms: Allocated to conventional vitamin C (n= 22)
Dietary Supplement: placebo — The intake placebo was taken daily in the morning and the evening for 28 days (7 days before surgery, on the day of surgery and twenty-one days after the surgical procedure).
  Arms: Allocated to placebo (n= 22)

SUMMARY:
Abstract:

Complex regional pain syndrome (CRPS) is a significant complication in operated osteoarticular pathology and may adversely affect patient's quality of life. Vitamin C is an anti-oxidant and a neuro-modulating agent. Intake of vitamin C appears to be the only preventative factor. The objective of this study seeks to assess the effectiveness of liposomal conditioning of vitamin-C in reducing CRPS and to show evidence that it is more effective than taking vitamin C in its usual form.

DETAILED DESCRIPTION:
Methods:

Three series of patients undergone for identical pathologies the same surgery performed in the same centre by a single surgeon using the same operative techniques and the same implants. The first group took vitamin C in liposomal form. The second one took classical vitamin C tablets while the third one received placebo pills. Comparison was made between both groups which were identical in number and were the same average age. Results were compared and analysed at the end of one-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Female, Age > 18 years
* The woman of childbearing age - if applicable - must have a negative urine pregnancy test result and must agree to use adequate contraception (hormonal or barrier contraception method, or abstinence) during the study and one month later)
* Consenting patient
* Agrees to maintain the current level of physical activity throughout the study.
* Agrees to avoid vitamins and supplements for 30 days before enrolment and during the study.
* Avoid nutritious yeasts, whey protein, energy drinks, pomegranate, pomegranate juice, grapefruit, grapefruit juice and alcohol 7 days before enrolment and during the study
* Willingness and ability to comply with scheduled visits, cellular phone calls, treatment plans, laboratory tests and completion of other study procedures specified in the protocol.

Exclusion Criteria:

* Pregnant, breastfeeding or considering pregnancy during the trial
* Diabetic women
* No renal lithiasis
* No deficiency Glucose-6-phosphate dehydrogenase
* Unstable medical conditions
* Immunocompromised persons such as subjects who have undergone organ transplantation
* Subjects who planned surgery during the clinical study
* History of blood disorders / bleeding
* Alcohol abuse (> 2 standard alcoholic beverages per day) or drug addiction in the last 6 months
* Participation in a clinical research trial within 30 days of randomization
* Allergy or sensitivity to the product during the clinical study.
* Persons who have a cognitive impairment and/or are unable to give an informed opinion.
* Any other condition that, in the opinion of the physician, could affect the subject and lead to the successful completion of the study, action or pose a significant risk to the subject.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2019-06-19 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 5 years
Access Criteria: Information will be given after approval.

REFERENCES:
- [Background] Camelot C, Ramare S, Lemoine J, Saillant G. [Orthopedic treatment of fractures of the lower extremity of the radius by the Judet technique. Anatomic results in function of the type of lesion: apropos of 280 cases]. Rev Chir Orthop Reparatrice Appar Mot. 1998 Apr;84(2):124-35. French. PMID 9775056
- [Background] van der Laan L, Kapitein PJ, Oyen WJ, Verhofstad AA, Hendriks T, Goris RJ. A novel animal model to evaluate oxygen derived free radical damage in soft tissue. Free Radic Res. 1997 Apr;26(4):363-72. doi: 10.3109/10715769709097816. PMID 9167941
- [Background] Matsuda T, Tanaka H, Shimazaki S, Matsuda H, Abcarian H, Reyes H, Hanumadass M. High-dose vitamin C therapy for extensive deep dermal burns. Burns. 1992 Apr;18(2):127-31. doi: 10.1016/0305-4179(92)90009-j. PMID 1590927
- [Background] Zollinger PE, Tuinebreijer WE, Kreis RW, Breederveld RS. Effect of vitamin C on frequency of reflex sympathetic dystrophy in wrist fractures: a randomised trial. Lancet. 1999 Dec 11;354(9195):2025-8. doi: 10.1016/S0140-6736(99)03059-7. PMID 10636366
- [Background] Cazeneuve JF, Leborgne JM, Kermad K, Hassan Y. [Vitamin C and prevention of reflex sympathetic dystrophy following surgical management of distal radius fractures]. Acta Orthop Belg. 2002 Dec;68(5):481-4. French. PMID 12584978
- [Background] Aim F, Klouche S, Frison A, Bauer T, Hardy P. Efficacy of vitamin C in preventing complex regional pain syndrome after wrist fracture: A systematic review and meta-analysis. Orthop Traumatol Surg Res. 2017 May;103(3):465-470. doi: 10.1016/j.otsr.2016.12.021. Epub 2017 Mar 4. PMID 28274883
- [Background] Harden NR, Bruehl S, Perez RSGM, Birklein F, Marinus J, Maihofner C, Lubenow T, Buvanendran A, Mackey S, Graciosa J, Mogilevski M, Ramsden C, Chont M, Vatine JJ. Validation of proposed diagnostic criteria (the "Budapest Criteria") for Complex Regional Pain Syndrome. Pain. 2010 Aug;150(2):268-274. doi: 10.1016/j.pain.2010.04.030. Epub 2010 May 20. PMID 20493633
- [Background] Elhusseiny KM, Abd-Elhay FA, Kamel MG, Abd El Hamid Hassan HH, El Tanany HHM, Hieu TH, Tieu TM, Low SK, Hou V, Dibas M, Huy NT. Examined and positive lymph nodes counts and lymph nodes ratio are associated with survival in major salivary gland cancer. Head Neck. 2019 Aug;41(8):2625-2635. doi: 10.1002/hed.25742. Epub 2019 Mar 23. PMID 30905082
- [Background] Abd-Elhay FA, Elhusseiny KM, Kamel MG, Low SK, Sang TK, Mehyar GM, Nhat Minh LH, Hashan MR, Huy NT. Negative Lymph Node Count and Lymph Node Ratio Are Associated With Survival in Male Breast Cancer. Clin Breast Cancer. 2018 Dec;18(6):e1293-e1310. doi: 10.1016/j.clbc.2018.07.003. Epub 2018 Jul 7. PMID 30093263
- [Background] de Thomasson E, Rouvreau P, Piriou P, Fitoussi F, Boury G, Judet T. [Orthopaedic treatment of colles' fractures according to judet's method]. Eur J Orthop Surg Traumatol. 1995 Dec;5(2):87-92. doi: 10.1007/BF02716246. French. PMID 24193325
- [Background] Roumen RM, Hesp WL, Bruggink ED. Unstable Colles' fractures in elderly patients. A randomised trial of external fixation for redisplacement. J Bone Joint Surg Br. 1991 Mar;73(2):307-11. doi: 10.1302/0301-620X.73B2.2005162.
- [Background] Cooney WP 3rd, Dobyns JH, Linscheid RL. Complications of Colles' fractures. J Bone Joint Surg Am. 1980;62(4):613-9. PMID 6155380
- [Background] Stanton-Hicks M, Janig W, Hassenbusch S, Haddox JD, Boas R, Wilson P. Reflex sympathetic dystrophy: changing concepts and taxonomy. Pain. 1995 Oct;63(1):127-133. doi: 10.1016/0304-3959(95)00110-E. PMID 8577483
- [Background] van der Laan L, ter Laak HJ, Gabreels-Festen A, Gabreels F, Goris RJ. Complex regional pain syndrome type I (RSD): pathology of skeletal muscle and peripheral nerve. Neurology. 1998 Jul;51(1):20-5. doi: 10.1212/wnl.51.1.20. PMID 9674773
- [Background] Oyen WJG, Arntz IE, Claessens RAMJ, Van der Meer JWM, Corstens FHM, Goris JAR. Reflex sympathetic dystrophy of the hand: an excessive inflammatory response? Pain. 1993 Nov;55(2):151-157. doi: 10.1016/0304-3959(93)90144-E. PMID 8309706
- [Background] Tanaka H, Broaderick P, Shimazaki S, Matsuda H, Hansalia H, Hanumadass M, Reyes H, Matsuda T. How long do we need to give antioxidant therapy during resuscitation when its administration is delayed for two hours? J Burn Care Rehabil. 1992 Sep-Oct;13(5):567-72. doi: 10.1097/00004630-199209000-00010. PMID 1452591
- [Background] Zollinger PE, Tuinebreijer WE, Breederveld RS, Kreis RW. Can vitamin C prevent complex regional pain syndrome in patients with wrist fractures? A randomized, controlled, multicenter dose-response study. J Bone Joint Surg Am. 2007 Jul;89(7):1424-31. doi: 10.2106/JBJS.F.01147. PMID 17606778
- [Background] Ekrol I, Duckworth AD, Ralston SH, Court-Brown CM, McQueen MM. The influence of vitamin C on the outcome of distal radial fractures: a double-blind, randomized controlled trial. J Bone Joint Surg Am. 2014 Sep 3;96(17):1451-9. doi: 10.2106/JBJS.M.00268. PMID 25187584
- [Background] Reuben SS. Preventing the development of complex regional pain syndrome after surgery. Anesthesiology. 2004 Nov;101(5):1215-24. doi: 10.1097/00000542-200411000-00023. No abstract available. PMID 15505459
- [Background] Besse JL, Gadeyne S, Galand-Desme S, Lerat JL, Moyen B. Effect of vitamin C on prevention of complex regional pain syndrome type I in foot and ankle surgery. Foot Ankle Surg. 2009;15(4):179-82. doi: 10.1016/j.fas.2009.02.002. Epub 2009 Apr 5. PMID 19840748
- [Background] Shibuya N, Humphers JM, Agarwal MR, Jupiter DC. Efficacy and safety of high-dose vitamin C on complex regional pain syndrome in extremity trauma and surgery--systematic review and meta-analysis. J Foot Ankle Surg. 2013 Jan-Feb;52(1):62-6. doi: 10.1053/j.jfas.2012.08.003. Epub 2012 Sep 15. PMID 22985495
- [Background] Sabesan VJ, Shahriar R, Petersen-Fitts GR, Whaley JD, Bou-Akl T, Sweet M, Milia M. A prospective randomized controlled trial to identify the optimal postoperative pain management in shoulder arthroplasty: liposomal bupivacaine versus continuous interscalene catheter. J Shoulder Elbow Surg. 2017 Oct;26(10):1810-1817. doi: 10.1016/j.jse.2017.06.044. Epub 2017 Aug 24. PMID 28844420

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All of 66 participants met the inclusion criteria and were randomised to treatment.
Groups:
- Allocated to Conventional Vitamin C (n= 22): Participant intake of traditional vitamin C with a daily intake of 500 mg in the morning and evening for 28 days (starting 7 days before the operative procedure, on the day of the surgery and ending twenty-one days after surgery).
- Allocated to Liposomal Vitamin C (n= 22): Participant intake of liposomal vitamin C at 500 mg, in the morning and evening, one week before surgery, one during the day of surgery and lastly, during the first 21 post operation days.
- Allocated to Placebo (n= 22): Participant intake placebo was taken daily in the morning and the evening for 28 days (7 days before surgery, on the day of surgery and twenty-one days after the surgical procedure).
Period: Overall Study
Arm/Group | Allocated to Conventional Vitamin C (n= 22) | Allocated to Liposomal Vitamin C (n= 22) | Allocated to Placebo (n= 22)
Started | 22 | 22 | 22
Completed | 22 | 22 | 22
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allocated to Conventional Vitamin C (n= 22) | Allocated to Liposomal Vitamin C (n= 22) | Allocated to Placebo (n= 22) | Total
Number analyzed (Participants) | 22 | 22 | 22 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (9.46) | 44 (9.64) | 43.77 (9.29) | 43.9 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 22 | 66
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  France | 22 | 22 | 22 | 66
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 21.75 (2.1) | 21.57 (2.07) | 21.75 (1.98) | 21.69 (2)
Surgery (%) [Count of Participants; unit: Participants]
  ACL(anterior cruciate ligament) | 5 | 5 | 5 | 15
  TKA = total knee arthroplasty | 6 | 6 | 6 | 18
  UKA = unicompartmental knee arthroplasty | 6 | 6 | 6 | 18
  ATO = anterior tibial osteotomy | 5 | 5 | 5 | 15
Complications (%) [Count of Participants; unit: Participants]
  None | 10 | 12 | 10 | 32
  Laxity | 1 | 1 | 1 | 3
  Pain | 6 | 2 | 6 | 14
  Stiffness | 2 | 2 | 2 | 6
  Patella Pain | 1 | 2 | 1 | 4
  Unimproved | 2 | 3 | 2 | 7
Scintigraphy (%) [Count of Participants; unit: Participants]
  Negative | 7 | 9 | 6 | 22
  Not made | 10 | 13 | 10 | 33
  CRPS = complex regional pain syndrome. | 5 | 0 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Operated for Complex Regional Pain Syndrome Who Had Transposition of Anterior Tibial Tuberosity
Description: We take an x-ray of the knee then we calculate of the Index of Caton and Deschamps AT / AP which must be close to 1 cm (from the upper edge to the lower edge of the patella which must be equal to the distance between the tip of the patella and anterior tibial tuberosity) to be interpreted as a transposed tuberosity.
Time Frame: After one-year of follow-up
Population: Among 15 patients who had transposition of anterior tibial tuberosity, results shows the number of cases operated for complex regional pain syndrome (CRPS).
Measure: Number; unit: participants
Arm/Group | Allocated to Conventional Vitamin C (n= 22) | Allocated to Liposomal Vitamin C (n= 22) | Allocated to Placebo (n= 22)
Number analyzed (Participants) | 5 | 5 | 5
participants | 1 | 0 | 2

2. Primary Outcome: Number of Participants Operated for Complex Regional Pain Syndrome Who Had Ligamentoplasty ACL According to Kenneth-Jones
Description: Radiographs of the knee in monopodial support at 30° flexion (schuss) were taken. Measurement analysis of the translation of the tibia relative to the femur which must be close to 0 cm for the patient to be positive for the outcome.
Time Frame: After one-year follow-up
Population: Among 15 patients who had Ligamentoplasty (ACL) according to Kenneth-Jones, results shows the number of cases operated for complex regional pain syndrome (CRPS)
Measure: Number; unit: participants
Arm/Group | Allocated to Conventional Vitamin C (n= 22) | Allocated to Liposomal Vitamin C (n= 22) | Allocated to Placebo (n= 22)
Number analyzed (Participants) | 5 | 5 | 5
participants | 1 | 0 | 0

3. Primary Outcome: Number of Participants Operated for Complex Regional Pain Syndrome Who Had Internal Unicompartmental Arthroplasty for Centralized Arthritis
Description: Radiographs of the knee in Schuss with an external decoaptation which must be close to 0 cm and a pan gono gram standing from the front
Time Frame: After one-year follow-up
Population: Among 18 patients who had Internal unicompartmental arthroplasty for centralized arthritis, results shows the number of cases operated for complex regional pain syndrome (CRPS)
Measure: Number; unit: participants
Arm/Group | Allocated to Conventional Vitamin C (n= 22) | Allocated to Liposomal Vitamin C (n= 22) | Allocated to Placebo (n= 22)
Number analyzed (Participants) | 6 | 6 | 6
participants | 0 | 0 | 0

4. Primary Outcome: Number of Participants Operated for Complex Regional Pain Syndrome Who Had Total Knee Arthroplasty for Eccentric Arthritis
Description: X-rays of the knee and Schuss profile with an internal and external decoaptation which must be close to 0 cm with pan gonogram standing from the front (x-rays of the long axes of the pelvis of the ankles with measurement of the HKA axes on the prosthesis side and on the non-side operated which must be close to 180°) to have eccentric arthritis.
Time Frame: After one-year follow-up
Population: Among 18 patients who had Total knee arthroplasty for eccentric arthritis, results shows the number of cases operated for complex regional pain syndrome (CRPS)
Measure: Number; unit: participants
Arm/Group | Allocated to Conventional Vitamin C (n= 22) | Allocated to Liposomal Vitamin C (n= 22) | Allocated to Placebo (n= 22)
Number analyzed (Participants) | 6 | 6 | 6
participants | 1 | 0 | 2

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | Allocated to Conventional Vitamin C (n= 22) | Allocated to Liposomal Vitamin C (n= 22) | Allocated to Placebo (n= 22)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT04204200/Prot_SAP_000.pdf